CLINICAL TRIAL: NCT06405230
Title: A Pilot/Exploratory Translational Study to Evaluate Response to Dostarlimab and Pembrolizumab in Extracellular Vesicles (EVs) or Patient-derived Organoids (PDOs) and by Zirconium-89 Labelled Programmed Death Ligand 1 Positron Emission Tomography in Participants With Recurrent Non-small Cell Lung Cancer
Brief Title: Evaluation of Programmed Death Ligand 1 (PDL1) Response to Treatment in Extracellular Vesicles (EVs), Patient-derived Organoid (PDOs)s and Immune-marker Positron Emission Tomography (PET) Scanning in Non-small Cell Lung Cancer (NSCLC)
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 221861
Record Dates: First submitted 2024-04-18; First posted 2024-05-08 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer, Non-Small Cell
Keywords: Non-small cell lung cancer; Pembrolizumab; Dostarlimab; Platinum-based chemotherapy doublet; Programmed death ligand 1; Positron emission tomography; Extracellular Vesicles; Organoids; Artificial intelligence; Machine learning
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; dostarlimab; Pemetrexed; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab ± Platinum-based chemotherapy doublet (PBCD) (Experimental): Participants will receive pembrolizumab with or without PBCD.
  Interventions: Biological: Pembrolizumab; Drug: Pemetrexed+ (carboplatin or cisplatin)
- Dostarlimab ± PBCD (Experimental): Participants will receive dostarlimab with or without PBCD.
  Interventions: Biological: Dostarlimab; Drug: Pemetrexed+ (carboplatin or cisplatin)

INTERVENTIONS:
Biological: Pembrolizumab — Pembrolizumab will be administered.
  Arms: Pembrolizumab ± Platinum-based chemotherapy doublet (PBCD)
Biological: Dostarlimab — Dostarlimab will be administered.
  Arms: Dostarlimab ± PBCD
Drug: Pemetrexed+ (carboplatin or cisplatin) — PBCD consisting of pemetrexed+ (carboplatin or cisplatin) will be administered.

SUMMARY:
The goal of this clinical trial is to investigate the utility of biomarker tools Extracellular Vesicles (EVs), Patient-derived organoid (PDOs), and PDL1 PET imaging for predicting how participants with recurrent NSCLC respond to standard of care treatment in the advanced/metastatic stages.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically- or cytologically documented NSCLC who present with recurrent advanced or metastatic disease after initial diagnosis of Stage 1-3 lung cancer
* Participants must have been initially diagnosed with operable Stage 1-3 NSCLC and received curative resection ± (neo) adjuvant treatment
* Identifiable PDL1 status prior to randomisation
* Participants must have biopsy-confirmed recurrence of their initial NSCLC with advanced/metastatic presentation
* Has at least 1 measurable (target) lesion per Response Evaluation Criteria in Solid Tumours (RECIST) version (v) 1.1 by Computed tomography (CT) or magnetic resonance imaging (MRI). Measurable lesions that have been previously irradiated are not considered measurable and cannot be target lesions
* Participants must be deemed by investigator to be appropriate to receive 1L systemic therapy (i.e., anti-PD1 ± PBCD)
* Participants must have had tissue submitted for attempted PDO generation. (Note: patients deemed to have successfully established paired 1o PDO [from the tumour resection at time of diagnosis]are those whose PDO cultures have been passaged 2 times, with a reasonable proliferation rate. This designation can be made prior to or during trial participation. A KCL biobank pathologist will confirm the PDO's representation of clinical tumour tissue sample at the time of multiomic analysis).
* Participants with known human immunodeficiency virus (HIV) infection are allowed with the following requirements:

  1. Documented evidence of plasma HIV-1 ribonucleic acid (RNA) persistently <50 copies per millilitre (c/mL) ≤3 months prior to and at Screening. In the >3 to 12 months prior to Screening, plasma HIV-1 RNA consistently <50 c/mL required; if single increases ≥50 c/mL occurred, they cannot have been persistent nor associated with antiretroviral resistance per investigator assessment
  2. cluster of differentiation 4 (CD4) cell count >350 cells per cubic millimetre (cells/mm^3) over past 12 months and at Screening (and no measurement ≤350 cells/mm3 during that time period)
  3. Must be on an uninterrupted combination antiretroviral therapy regimen for at least 3 months prior to Screening, with combination antiretroviral therapy regimen consistent with locally recommended guidelines
  4. Participants with history of Centres for Disease Control and Prevention (CDC) Stage 3 acquired immunodeficiency syndrome (AIDS)-defining disease are allowed if AIDS-defining disease has been treated and cured or is stable for ≥3 months prior to study entry. Cutaneous Kaposi's sarcoma not requiring systemic therapy is allowed
  5. No history of HIV-associated non-Hodgkin lymphoma ≤5 years prior to study entry
  6. No treatment with an HIV-1 immunotherapeutic vaccine within 90 days of Screening
* Fresh tumour biopsy (taken as part of disease recurrence evaluation) is a requirement, provided that a biopsy procedure is technically feasible and the procedure is not associated with unacceptable clinical risk. If fresh biopsy sample is not available, an archival sample may be used
* Has an Eastern Cooperative Oncology Group Performance Status (ECOG PS) of 0 to 2
* Has adequate organ function per the investigator

Exclusion Criteria:

* Mixed lung carcinoma (small cell carcinoma and NSCLC), small cell carcinoma, large cell neuroendocrine carcinoma, sarcomatoid carcinoma, or any other histologies that would not benefit from anti-PD1 ± PBCD. If a potential participant has histology other than squamous cell or adenocarcinoma (e.g., mixed histology that is predominantly NSCLC, large cell without neuroendocrine features) but is deemed appropriate for treatment with anti-PD1 ± PBCD, they may be eligible pending discussion with the sponsor.
* For participants who received adjuvant therapy that included anti-PD(L)1 Checkpoint inhibitor (CPI) following surgical resection, their last dose of anti-PD(L)1 was <6 months from the date of first 89Zr-durvalumab-PET tracer injection
* Participant has known central nervous system (CNS) metastases and/or carcinomatous meningitis that per investigator puts the participant at prohibitive risk to enrol in study
* Participant has a known additional malignancy that progressed or required active treatment within the last 2 years. Participant with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with assessments of the study may be included only after discussion with the Medical Monitor
* Participant is considered a poor medical risk by the investigator due to a serious, uncontrolled medical disorder, non-malignant systemic disease or active infection requiring systemic therapy. Specific examples include, but are not limited to, active, non-infectious pneumonitis; uncontrolled chronic obstructive pulmonary disease; uncontrolled ventricular arrhythmia; recent (within 90 days) myocardial infarction; uncontrolled major seizure disorder; unstable spinal cord compression; superior vena cava syndrome; or any psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the study (including obtaining informed consent)
* Participant is pregnant or breastfeeding or expecting to conceive children within the projected duration of the study, starting with the Screening Visit through 150 days after the last dose of study treatment
* Participant has a diagnosed immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy that per investigator puts the participant at prohibitive risk to enrol in the study
* Participant has an active HIV infection that per investigator puts the participant at prohibitive risk to enrol in study
* Participant has tested positive for the presence of hepatitis B surface antigen and/or Hepatitis B virus (HBV) core antibody or has a positive hepatitis C antibody test result at Screening or within 3 months prior to first dose of anti-cancer treatment
* Participant has an active autoimmune disease that has required systemic treatment (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy up to 5 milligrams (mg) prednisone or equivalent for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment. Use of inhaled steroids, topical steroids, local injection of steroids, and steroid eye drops are allowed
* Participant has history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan that per investigator and medical monitor puts the participant at prohibitive risk to enrol in study
* Participant is currently participating and receiving study therapy or has participated in a study of an investigational agent and received investigational therapy or used an investigational device within 4 weeks prior to the first dose of study drug
* Has cirrhosis or current unstable liver or biliary disease per investigator assessment defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, oesophageal/gastric varices, or persistent jaundice
* Participant has not recovered adequately (≤ Grade 1) per investigator from AEs and/or complications from any major surgery prior to starting therapy
* Participant has received a vaccine other than a vaccine against Severe acute respiratory syndrome coronavirus disease 19 (SARS-CoV-2) infection (COVID-19) within 7 days of planned start of study therapy. The use of all COVID-19 vaccines is allowed, with the exception of COVID-19 vaccines using the recombinant adenoviral vector platform within 30 days of planned start of study therapy. If a COVID-19 vaccine using this platform is to be administered within 30 days of planned start of study therapy, this must first be discussed with and approved by the sponsor's medical monitor
* Participant has received any form of anti-cancer therapy (e.g., chemotherapy, radiation, immunotherapy) for lung cancer recurrence after initial surgery
* Is receiving any additional anticancer post-surgery±(neo) adjuvant therapy or experimental therapy. No other experimental therapies (including but not limited to chemotherapy, radiation, hormonal treatment, antibody therapy, immunotherapy, gene therapy, vaccine therapy, or other experimental drugs) of any kind are permitted while the participant is receiving study intervention
* NSCLC with known sensitizing EGFR mutations, Anaplastic lymphoma kinase (ALK) translocations, or c-ros oncogene 1 (ROS1) mutations from resected tissue at the time of initially surgery and/or tissue biopsy at the time of screening
* Has a history of severe allergic and/or anaphylactic reactions to chimeric, human or humanized antibodies, fusion proteins, or known allergies to pembrolizumab, dostarlimab, durvalumab, or their excipients
* Symptomatic herpes zoster within 3 months prior to screening
* Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, chest X-rays (posterior anterior and lateral), and TB testing: either a positive Tuberculin skin test (TST) (defined as a skin induration ≥5 millimetres [mm] at 48 to 72 hours, regardless of Bacillus Calmette-Guerin or other vaccination history) or a positive (not indeterminate) TB test such as QuantiFERON-TB Gold Plus test
* QT interval corrected for heart rate according to Fridericia's formula (QTc) >450 milliseconds (msec) or QTc >480 msec in participants with bundle branch block

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-30 (Actual); Primary Completion 2028-08-07 (Estimated); Study Completion 2029-10-10 (Estimated)

PRIMARY OUTCOMES:
Spearman's rank correlation coefficient between treatment-induced PDL1 modulation in, 1o PDOs and/or extracellular vesicles (EVs) and PET after treatment | Up to approximately 29 months
  The primary endpoint is the correlation between "treatment-induced change in PDL1 in PDOs which will be evaluated as the ratio of PDL1 positive cells before and after treatment using flow cytometry and multiplex immunofluorescence analysis" AND/OR "treatment-induced change in PDL1 in EVs which will be evaluated as the ratio of PDL1 positive cells before and after treatment using flow cytometry and multiplex immunofluorescence analysis" and "changes in PET which will be evaluated as the percentage difference in PDL1-PET standard uptake volume (SUV) uptake in lesions from the baseline to on-treatment" using the formula for Spearman's rank correlation coefficient. The Spearmans rank correlation coefficient can take values from +1 to -1 where a value of +1 indicates a perfect positive association, a value of 0 indicates no association and a value of -1 indicates a perfect negative association.

SECONDARY OUTCOMES:
Spearman's rank correlation coefficient between treatment-induced PDL1 modulation in 1o PDOs and tumour response to anti- Programmed death 1 (PD1) based first line (1L) advanced/metastatic NSCLC treatment | Up to approximately 34.5 months
  The secondary endpoint is the correlation between "treatment-induced change in PDL1 in PDOs which will be evaluated as the ratio of PDL1 positive cells before and after treatment using flow cytometry and multiplex immunofluorescence analysis" AND "tumor response rate which will be assessed based on RECIST v1.1 per investigator assessment" using the formula for Spearman's rank correlation coefficient. The Spearmans rank correlation coefficient can take values from +1 to -1 where a value of +1 indicates a perfect positive association, a value of 0 indicates no association and a value of -1 indicates a perfect negative association.
Spearman's rank correlation coefficient between treatment-induced PDL1 modulation in EVs and tumour response to anti- Programmed death 1 (PD1) based first line (1L) advanced/metastatic NSCLC treatment | Up to approximately 34.5 months
  The secondary endpoint is the correlation between "treatment-induced change in PDL1 in EVs which will be evaluated as the ratio of PDL1 positive cells before and after treatment using flow cytometry and multiplex immunofluorescence analysis" AND "tumor response rate which will be assessed based on RECIST v1.1 per investigator assessment" using the formula for Spearman's rank correlation coefficient. The Spearmans rank correlation coefficient can take values from +1 to -1 where a value of +1 indicates a perfect positive association, a value of 0 indicates no association and a value of -1 indicates a perfect negative association.
Spearman's rank correlation coefficient between treatment-induced PDL1 modulation by PET and radiological tumour response to anti-PD1 based 1L advanced/metastatic NSCLC treatment | Up to approximately 34.5 months
  The secondary endpoint is the correlation between "changes in PET which will be evaluated as the percentage difference in PDL1-PET standard uptake volume (SUV) uptake in lesions from the baseline to on-treatment" AND "tumor response rate which will be assessed based on RECIST v1.1 per investigator assessment" using the formula for Spearman's rank correlation coefficient. The Spearmans rank correlation coefficient can take values from +1 to -1 where a value of +1 indicates a perfect positive association, a value of 0 indicates no association and a value of -1 indicates a perfect negative association.
Number of participants with adverse events (AEs) and serious adverse events (SAEs) following Zirconium-89 (89Zr-durvalumab)-PET radiotracer injection | Up to Week 4
Number of participants with treatment emergent AEs (TEAEs), immune-related AEs, and SAEs by severity | Up to approximately 34.5 months
Number of participants with TEAEs or SAEs, leading to dose delays, withdrawals, or death | Up to approximately 34.5 months
Number of participants with clinically significant changes in laboratory, vital signs, and safety assessment parameters | Up to approximately 34.5 months

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/